CLINICAL TRIAL: NCT05085015
Title: Effects of Exercise Training on Cardiometabolic Risk Factors and Functional Capacity in Individuals Undergoing Bariatric Surgery
Brief Title: Effects of Exercise Training in Individuals Undergoing Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Eastern Mediterranean University (Other)
Responsible Party: Principal Investigator, Hayriye Tomaç, Principal Investigator specialist physiotherapist, Eastern Mediterranean University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Unique Protocol ID: 2021-0071
Record Dates: First submitted 2021-05-24; First posted 2021-10-20 (Actual); Last update posted 2023-01-18 (Actual); Status verified 2023-01

CONDITIONS: Obesity
Keywords: Bariatrics; Obesity; Bariatric Surgery
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Functional Exercise Training Group (Experimental): A program including stretching, aerobics, strengthening and balance training will be implemented under the supervision of a physiotherapist with the instructions of the physiotherapist.They will apply a total of 24 sessions of exercise program for 60-80 minutes, 3 days a week, 8 weeks.
  Interventions: Other: Functional Exercise Training Group
- Home Exercise Training Group (Experimental): Individuals in the home exercise training program will be asked to follow the program in accordance with the home exercise brochure given for 8 weeks, 3 days a week. The program will include stretching, aerobics, strengthening and balance training. The home exercise program will consist of a brochure prepared from a program similar to a functional exercise program.
  Interventions: Other: Home Exercise Training Group

INTERVENTIONS:
Other: Functional Exercise Training Group — Training will start with Stretching Training and end with stretching training. Stretching exercises targeting actively applied shoulder girdle, chest, neck, trunk, hip, front and back leg and ankle muscle groups will be given. Afterwards, it will be continued with Aerobic Exercise Training. The training will be given on the treadmill "Treadmill Technogym". Afterwards, it will be continued with Strengthening Training. Strength training will consist of a strengthening program that includes the lower extremity, upper extremity, trunk and core region. Elastic bands will be used in the training. Then, balance training will be given at the end.
  Arms: Functional Exercise Training Group
Other: Home Exercise Training Group — Training will start with Stretching Training and end with stretching training. Stretching exercises targeting actively applied shoulder girdle, chest, neck, trunk, hip, front and back leg and ankle muscle groups will be given. Afterwards, it will be continued with Aerobic Exercise Training. They will walk at least 30 minutes, 3 days a week for 8 weeks at outdoor. Afterwards, it will be continued with Strengthening Training. Strength training will consist of a strengthening program that includes the lower extremity, upper extremity, trunk and core region. Elastic bands will be used in the training. Then, balance training will be given at the end.
  Arms: Home Exercise Training Group

SUMMARY:
The subject of the research; Effects of exercise training on cardiometabolic risk factors and functional capacity in individuals undergoing bariatric surgery.

Purpose of the research; Cardiometabolic risk factors, body composition, muscle strength and endurance, posture, foot sense, physical exercise capacity, balance, pain, exercise benefits - barriers, exercise self-efficacy, exercise beliefs, to evaluate the effects on body esteem, body image and quality of life.

Method of Research:

Post-surgical interventions are important in individuals who have undergone bariatric surgery. Intervention programs that include exercise, encourage the change in the lifestyle of individuals, effectively and accurately reduce post-surgical obesity. Functional Exercise Training, which can also be used for obesity treatment, consists of stretching, aerobics, strengthening and balance training. Therefore, it has a positive effect on body systems. In addition, Home Exercise Training can be used within the scope of obesity treatment. Exercise is one of the alternative methods by providing the adaptation of the individual to the exercise. Socio-demographic and physical characteristics of individuals will be recorded. Laboratory tests will be ordered for cardiometabolic risk factors. Body composition will be determined by Tanita brand body analysis monitor (MC-780MA). Posture will be evaluated by photogrammetry technique. Muscle strength assessment will be evaluated by leg, back and hand dynamometer instrument, muscle endurance tests, sensory assessment by foot sense assessment, physical capacity with physical exercise capacity tests, balance static and dynamic balance tests and pain questionnaire. Exercise benefits-barriers will be assessed by Exercise Benefits Barriers Scale, exercise self-efficacy by Exercise Self-Efficacy Scale. Exercise beliefs will also be questioned with a questionnaire. Self-esteem will be evaluated for all groups before and after treatment. The self respect will be evaluated by using the Rosenberg Self-Esteem Scale, body image with the Body Image Scale, with the quality of life using the Obesity-Specific Quality of Life Scale.The training will be carried out 3 days a week for 8 weeks, approximately 1 hour. Sufficient number of assessments and exercises will be used for individuals to become familiar with the equipment and training protocol.

DETAILED DESCRIPTION:
Obesity is defined as abnormal or excessive fat accumulation in the body to the extent that it disrupts health. The prevalence of obesity is increasing day by day in developed and developing countries. While 600 million of the world population were obese in 2014, this situation reached 700 million in 2015, and when the trend continues in the same way, it is thought that more than 3 billion people will have overweight or obesity in 2030. Therefore, the worldwide prevalence of morbid obesity will increase rapidly. Obesity is a risk factor especially for cardiovascular disease and causes an increase in mortality and morbidity with the central accumulation of adipose tissues. It affects the muscle, liver, subcutaneous and intra-abdominal regions, especially due to intraabdominal and / or visceral fat. As a result, cardiometabolic complications occur, as it causes physical inactivity, muscle strength and endurance are affected, posture is affected, physical performance is affected, self-esteem, body image, health-related quality of life and exercise avoidance occur. It has been reported that approximately 91% of obese individuals complain of musculoskeletal pain, 69% of them have back pain and 58% have knee pain.

When the literature is examined, it is seen that conservative therapies such as nutrition, exercise and drug management are used intensively in the treatment of obesity, more invasive methods are more prominent today and bariatric surgery is preferred by many people. Studies emphasize that non-surgical methods fail to achieve permanent success compared to surgical methods. Obese individuals undergoing bariatric surgery have reported a large diet history that failed to stop weight gain, starting in adolescence. It has been reported that obese individuals experience higher levels of symptoms such as stress, anxiety, depression, food cravings and psychological effects such as lower self-esteem compared to normal weight individuals, and this situation continuously increases weight gain. For this reason, bariatric surgery has become increasingly common in the fight for effective weight loss. The postoperative process in which exercise and lifestyle changes are adopted after bariatric surgery is important. With the prominence of bariatric surgery in the studies performed, if weight loss management is not planned well after surgery, weight gain and complications occur after surgery, and it is seen that the effect of the surgery performed decreases. Weight recovery in this population also increases the likelihood of the return of obesity-related comorbidities. Insufficient physical activity and inadequate nutritional support after surgery cause sarcopenia. Therefore, it is an important anabolic stimulant for the prevention of muscle protein synthesis and sarcopenia formation, together with adequate nutritional support, together with early physical activity after surgery.

Increasing physical activity, exercise and lifestyle changes are important in maintaining the weight given during the postoperative period, reducing muscle loss and increasing fat burning. The purposes of exercise training given in the post-surgery period in obese individuals are to increase body fat mass loss, protect muscle mass, and improve physical and mental health. Although there are studies in which exercise training is important following bariatric surgery, there is insufficient evidence regarding the interventions of different exercise protocols. Finding the best exercise protocols, increasing body fat mass loss and preserving muscle mass is important as part of the post-surgical guideline. Studies have reported that physical exercise is a positive predictor of outcome after bariatric surgery. Intervention programs that include exercise are reported to effectively reduce obesity and comorbidity by encouraging individuals to change their lifestyle after such surgery. Studies have shown that exercise is considered an effective mediator for correcting insulin resistance, effectively reduces indicators of obesity such as body mass index (BMI) and body fat percentage, and reduced risk factors for cardiovascular diseases. Therefore, the main purpose of the study is to evaluate the effects of exercise training on cardiometabolic risk factors and functional capacity in individuals who have undergone bariatric surgery. There is no such exercise protocol study conducted in Cyprus. The investigators are of the opinion that the research is an interesting study in this respect.

Functional Exercise Training is a type of exercise that includes training for stretching, aerobics, strengthening and balance. Studies on obese individuals have reported a positive effect on body composition, functional capacity and quality of life.

Home Exercise Training, on the other hand, is one of the alternative methods of exercise that maximizes the sustainability of behavioral change by providing adaptation to exercise throughout life. It is an option that will increase an individual's physical activity compliance.

Evidence regarding the effectiveness of Functional Exercise Training and Home Exercise Training in Individuals Undergoing Bariatric Surgery is insufficient and it is necessary to know and clarify the differences create. It is necessary to clarify whether individuals continue the exercise in their daily lives and whether the continuity of the effects of the exercise should be addressed. In this context, the content and effects of the exercise programs to be applied to individuals who have undergone bariatric surgery are important in Cyprus for future multifactorial situations and may guide individuals.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 20-60 years,
* Those who have passed 1 month to 2 years after the operation,
* Lack of a regular exercise program for the last 6 months (3 and 20 minutes per week.

Exclusion Criteria:

* Uncontrollable Hypertension (systolic≥160, diastolic≤90 mmHg), Diabetes, Cancer and Cardiovascular Disease
* Those who have orthopedic, neurological or mental illnesses that prevent them from exercising
* Previous bariatric surgery
* Use of drugs that will affect body composition that will cause weight or energy expenditure
* Having vision, hearing and communication problems

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2021-12-10 (Actual); Primary Completion 2022-07-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | change from baseline at 8 weeks after the intervention
  Laboratory tests for the insulin resistance of the individuals will be obtained from the findings that are routinely requested and made by the doctor.
  For Insulin Resistance; Insulin resistance (HOMA-IR) test will be done by taking a blood test in the laboratory (Blood glucose taken after 8-10 hours of fasting and fasting insulin level will be multiplied by each other and divided by 405 and the insulin resistance level called HOMA-IR will be revealed.)

SECONDARY OUTCOMES:
Body Analysis Monitor | change from baseline at 8 weeks after the intervention
  Body composition will be evaluated with the Tanita brand body analysis monitor (MC-780MA).
  Tanita MC-780 is the multi frequency segmental body composition analyzer. This consists of a stand-alone unit where the subject has to step on barefoot and segmental values will be indicate by the end of the analysis on the digital screen.
Waist and hip circumference | change from baseline at 8 weeks after the intervention
  Waist and hip circumference will be measured. Waist / hip circumference ratio will be calculated.
Muscle Strength | change from baseline at 8 weeks after the intervention
  A leg and back dynamometer will be used to measure leg and back muscle strength. A hand dynamometer will be used for hand grip strength measurement. Both measurements will be made bilaterally.
Sorensen Test | change from baseline at 8 weeks after the intervention
  Sorensen Test; For trunk extensor muscle endurance
Trunk Flexor Muscle Endurance Test | change from baseline at 8 weeks after the intervention
  Trunk Flexor Muscle Endurance Test; For trunk flexor muscle endurance
Side Bridge Test (bilateral) | change from baseline at 8 weeks after the intervention
  Side Bridge Test (bilateral); For arm muscles providing lateral stability
Squat Test | change from baseline at 8 weeks after the intervention
  Squat Test; It will be applied for lower extremity muscle endurance
Posture Analysis | change from baseline at 8 weeks after the intervention
  Postural evaluation will be carried out using the photographic method. For this purpose, the photograph of the individual will be taken.
Foot Sense Assessment | change from baseline at 8 weeks after the intervention
  Foot sense will be evaluated by light touch and vibration sense measurement.
Time Up & Go Test | change from baseline at 8 weeks after the intervention
  This test is an objective, reliable and simple measure of balance and functional movement. It was developed by Podsiadlo and Richardson in 1991. The person will be asked to get up from a seat, walk 3 m, turn around, walk back to the seat and sit. It will be recorded how many seconds he finished the test.
Chair Sit & Go Test | change from baseline at 8 weeks after the intervention
  Subjects will be asked to sit in a chair with their hands crossed on their chests. They will be asked to sit up and stand up as fast as possible five times in a row. The test will be started in sitting position and the test will be terminated at the last take-off. The time in seconds will be kept. The test will be performed 2 times and the best score will be recorded.
Normal walking speed | change from baseline at 8 weeks after the intervention
  For normal walking, the person will be asked to walk a distance of 4 meters at a normal pace as in daily life, and the time to walk the 4 meters distance will be calculated in seconds. The test will be performed 2 times and the best score will be recorded.
Fast walking speed | change from baseline at 8 weeks after the intervention
  For fast walking, the person will be asked to walk a distance of 4 meters as fast as possible. The test will be done only once and the achieved grade will be recorded. Normal walking and fast walking speed will be recorded in m/s by dividing the distance by the recorded times.
One Foot Stand Test | change from baseline at 8 weeks after the intervention
  The time in seconds for individuals to stand on one leg, without shoes, by supporting their hands on their waists and bending their knees will be recorded. It will be done 2 times for each leg and the best score will be recorded.
Total physical capacity score | change from baseline at 8 weeks after the intervention
  As a result of the tests, the total physical capacity score will be obtained. Individuals '' Timed Up & Go Test (sec), Chair Sit & Go Test (sec), normal (m / sec) and fast walking speed (m / sec) and One Foot Stand Test (right / left average, sec) '' will be applied.
Balance | change from baseline at 8 weeks after the intervention
  Lower extremity Y balance test will be applied for Dynamic Balance. For Static Balance, eyes will be evaluated with open and closed eyes on one leg.
Short-Form Mcgill Pain Questionnaire | change from baseline at 8 weeks after the intervention
  Pain will be assessed by the Short-Form Mcgill Pain Questionnaire (SF-MAA). This form provides information about perceptual, sensory and severity components in pain perception. 15 descriptive adjectives (11 sensory and 4 affective) are used to determine the perception of pain. Descriptive adjectives in the pain perception of the cases are evaluated with a numerical value scale (0 = absent, 1 = mild, 2 = moderate, 3 = severe).
  In addition, ın this form have a visual analog scale of 10 cm is used to measure the pain intensity felt during the evaluation. They will be asked to indicate the pain they felt during the evaluation with an "X" mark on a 10 cm scale. According to this scale, a value of "0" indicates no pain, and "10" indicates the most severe pain. The distance between the marked point and the starting point is measured in cm.
Visual Analog Scale | change from baseline at 8 weeks after the intervention
  Visual analog scale of 10 cm is used to measure the pain intensity felt during the evaluation. They will be asked to indicate the pain they felt during the evaluation with an "X" mark on a 10 cm scale. According to this scale, a value of "0" indicates no pain, and "10" indicates the most severe pain. The distance between the marked point and the starting point is measured in cm.
  Accordingly, 0 means no pain, 10 means the most unbearable pain. Pain intensity increases as go to 10.
Exercise Benefits Barriers | change from baseline at 8 weeks after the intervention
  Exercise Benefits Barriers Scale will be evaluated to determine exercise benefit and obstacle perceptions of obese women.The scale is evaluated over the total score (min=24, max= 96). Higher scores indicate perceived greater exercise benefits and fewer exercise barriers.
Exercise Self-Efficacy | change from baseline at 8 weeks after the intervention
  With Exercise Self-Efficacy Scale, questions will be asked to measure the self-efficacy of obese women in exercising.A high total score from the scale indicates that the individual's self-efficacy perception is at a good level.
Exercise Beliefs | change from baseline at 8 weeks after the intervention
  Obese women will be asked to score according to the VAS scale to determine their physical activity beliefs. According to the VAS scale by asking the question "How important is physical activity for you?" It will be asked to mark on the scale. Accordingly, a score between 0 and 10 is made. 0 means no pain, 10 means the most unbearable pain. Pain intensity increases as go to 10
Self respect | change from baseline at 8 weeks after the intervention
  The Rosenberg Self-Esteem Scale will be used to evaluate the self-esteem of individuals.
  Low score in scale scoring means high self-esteem; a high score indicates low self-esteem.
  0-1 points as high self-esteem, 2-4 points as medium self-esteem, 5-6 points as low self-esteem
Body Image | change from baseline at 8 weeks after the intervention
  Body Image Scale will be used to evaluate the body image satisfaction level of individuals.
  The most positive statement gets 5 points, and the most negative statement gets 1 point. An increase in the total score obtained from the scale indicates an increase in satisfaction with one's body parts or function, and a decrease in a score indicates a decrease in satisfaction.
Life quality | change from baseline at 8 weeks after the intervention
  Obesity Specific Quality of Life Scale will be used to assess the quality of life.
  As the total score from the scale approaches 0, the quality of life decreases, and as it approaches 100, the quality of life increases.
Functional Exercise Capacity | change from baseline at 8 weeks after the intervention
  Six Minute Walk Test will be applied. The Six Minute Walk Test is a submaximal exercise test that evaluates exercise tolerance and exercise-related cardiorespiratory changes.
Lipid Profile | change from baseline at 8 weeks after the intervention
  Laboratory tests for the lipid profile of the individuals will be obtained from the findings that are routinely requested and made by the doctor. For this, blood findings will be taken in the analysis laboratory. For Lipid Profile; Triglycerides (TG), High-density lipoprotein cholesterol (HDL-C), Low-density lipoprotein cholesterol (LDL-C), Total cholesterol (TC), Glucose, Glycosylated Hemoglobin (HbA1c), C Reactive Protein (CRP) values will be checked in the results of blood tests. .
İnsulin Resistance | change from baseline at 8 weeks after the intervention
  Laboratory tests for the insulin resistance of the individuals will be obtained from the findings that are routinely requested and made by the doctor. For this, blood findings will be taken in the analysis laboratory. Insulin resistance test; The blood glucose taken after 8-10 hours of fasting will be multiplied by the fasting insulin level and divided by 405 and the insulin resistance level called HOMA-IR will appear. In this test, it will be checked as a result of blood tests to be taken in the laboratory.
Body weight | change from baseline at 8 weeks after the intervention
  Body weight will be evaluated in kg by measuring on a Tanita Brand body analysis monitor (MC-780MA).
Height | change from baseline at 8 weeks after the intervention
  Height is measured without shoes, heavy outer garments and hair ornaments. The back of the head, shoulder blades, buttocks and heels are touching the tape measure attached to the wall.The value in cm is taken.
Body mass index | change from baseline at 8 weeks after the intervention
  The Body Mass Index measurement will be obtained by dividing the weight in kilograms by the square of the height in meters (kg/m²) to arrive at a single reported value.

CONTACTS AND LOCATIONS:
Locations (1):
- Hayriye Tomaç, Famagusta, Cyprus

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code